CLINICAL TRIAL: NCT05457985
Title: Testing Adaptive Interventions to Improve Posttraumatic Stress Disorder (PTSD) Treatment Outcomes in Federally Qualified Health Centers
Brief Title: Testing Adaptive Interventions to Improve Posttraumatic Stress Disorder Treatment Outcomes in Federally Qualified Health Centers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Sripada, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00203165; 1R01MH125857-01A1 (NIH)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: PTSD
Keywords: Prolonged Exposure for Primary Care; Mobile device; Clinician Supported PTSD Coach App; PTSD symptoms; Prolonged Exposure/PE
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: All eligible participants will initially be randomized to one of the two first-stage options, either PE-PC or PTSD coach with clinician support. Participants that have experienced less than a 15-point reduction, have a PCL score of greater than 60 ("very severe"), or cannot be reached for assessment will be classified as slow responders and will be re-randomized to one of two second-stage tactics, either (a) continue in their first-stage treatment strategy, or (b) step up to full PE. Participants who have experienced at least a 15-point symptom reduction or have a PCL score of less than 29 will be classified as early responders and will step down to a lower intensity of their current treatment strategy (i.e., early responders will not be re-randomized).
Who Masked: Outcomes Assessor
Masking Description: The primary outcome, the Clinician-Administered PTSD Scale (CAP-5), will be administered by a blinded study team member.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Prolonged Exposure for Primary Care (PE-PC) then continue as early responder (Experimental): PE-PC consists of four weekly 30-minute sessions. At the 4th session or 9-week assessment point (whichever comes first), early responders will step down to every-other-week sessions for the duration of the second stage (for 8 weeks).
  Interventions: Behavioral: Prolonged Exposure for Primary Care (PE-PC)
- Clinician Supported (CS) PTSD Coach App then continue as early responder (Experimental): During the first stage of treatment, participants will receive four weekly clinician support sessions or 9 weeks (whichever occurs first). Early responders will be encouraged to continue app use but will discontinue clinician support sessions for the remaining 8 weeks.
  Interventions: Behavioral: Clinician Supported PTSD Coach App
- Prolonged Exposure for Primary Care (PE-PC) then full PE (Experimental): PE-PC consists of four weekly 30-minute sessions. At the 4th session or 9-week assessment point (whichever comes first), slow responders that are then randomized to full PE and will have sessions once a week for eight weeks. During these 60-minute sessions, participants will practice in vivo and imaginal exposure and continue these exposure exercises every day at home.
  Interventions: Behavioral: Prolonged Exposure for Primary Care (PE-PC); Behavioral: Full Prolonged Exposure
- Clinician Supported PTSD Coach App then full PE (Experimental): During the first stage of treatment, participants will receive four weekly clinician support sessions or 9 weeks (whichever occurs first), slow responders that are then randomized to full PE will have sessions once a week for eight weeks. During these 60 minute sessions, participants will practice in vivo and imaginal exposure and continue these exposure exercises every day at home.
  Interventions: Behavioral: Full Prolonged Exposure; Behavioral: Clinician Supported PTSD Coach App
- Prolonged Exposure for Primary Care (PE-PC) then continued PE-PC (Experimental): PE-PC consists of four weekly 30-minute sessions. At the 4th session or 9-week assessment point (whichever comes first), slow responders that are then randomized to continue with PE-PC (medium intensity) will continue weekly sessions for 8 weeks.
  Interventions: Behavioral: Prolonged Exposure for Primary Care (PE-PC)
- Clinician Supported PTSD Coach App then continued CS PTSD Coach App (Experimental): During the first stage of treatment, participants will receive four weekly clinician support sessions or 9 weeks (whichever occurs first), slow responders that are then randomized to continue this treatment will have the frequency reduced to twice monthly.
  Interventions: Behavioral: Clinician Supported PTSD Coach App

INTERVENTIONS:
Behavioral: Prolonged Exposure for Primary Care (PE-PC) — Treatment follows the standardized PE-PC manual and workbook.PE-PC consists of four weekly 30-minute sessions. In vivo and imaginal exposure are introduced at the first session and reviewed at Sessions 2-4. To conduct in vivo exposure, participants repeatedly and systematically approach objectively safe people, places, objects, and situations that they avoid because these stimuli remind them of their trauma. At the 4th session or 9-week assessment point (whichever comes first), early responders will step down to every-other-week sessions for the duration of the second stage.
  Arms: Prolonged Exposure for Primary Care (PE-PC) then continue as early responder; Prolonged Exposure for Primary Care (PE-PC) then continued PE-PC; Prolonged Exposure for Primary Care (PE-PC) then full PE
Behavioral: Full Prolonged Exposure — Treatment will follow the standardized PE manual. Participants will have 60 minute sessions once a week for eight weeks During these sessions, participants will practice in vivo, imaginal, and emotional exposure as well as continue these exposure exercises every day at home.
  Arms: Clinician Supported PTSD Coach App then full PE; Prolonged Exposure for Primary Care (PE-PC) then full PE
Behavioral: Clinician Supported PTSD Coach App — This is a brief psychotherapy that uses the PTSD Coach mobile app developed by the study team. The PTSD Coach app incorporates evidence-based assessment, psychoeducation, and cognitive behavioral therapy and self-management strategies that are customizable to the user.
  Arms: Clinician Supported (CS) PTSD Coach App then continue as early responder; Clinician Supported PTSD Coach App then continued CS PTSD Coach App; Clinician Supported PTSD Coach App then full PE

SUMMARY:
This trial is being completed to develop a stepped-care talk therapy model for patients with PTSD. Specifically, this study is testing whether beginning with one type of therapy is better than beginning with another type of therapy, and whether moving to a different therapy after four sessions is more helpful than staying with the same therapy, depending on how well it is working.

The central hypothesis is that beginning with a low- or medium-intensity PTSD intervention and then titrating intensity based on early indications of response will result in clinically significant PTSD symptom reduction with parsimony of resources.

ELIGIBILITY:
Inclusion Criteria:

* Receive care at a participating federally qualified health center (FQHC)
* Have a Posttraumatic Stress Disorder checklist (PCL-5) score greater or equal (≥) to 33
* Own a mobile device that can be used for the PTSD Coach App
* Have had psychotropic medication stability for at least 4 weeks

Exclusion Criteria:

* Severe cognitive impairment that in the judgment of the investigators makes it unlikely that the participant can adhere to the study regimen (as evidenced by confusion, inability to track discussion or answer questions, or other clear and significant indicators of cognitive impairment)
* High risk of suicide (defined as meeting criteria for Action Step 3 on the Participant Suicide Risk Screening form
* Severe alcohol or substance use disorder (moderate-severe alcohol use disorder on Alcohol Use Disorders Identification Test (AUDIT) (scores ≥ 15) or high risk on National Institute on Drug Abuse Quick Screen (scores ≥ 27))
* Active psychosis or unmanaged bipolar disorder
* Unstable housing
* Current engagement in a trauma-focused behavioral treatment (such as Prolonged Exposure or Cognitive Processing Therapy).
* Patients who do not speak English will be excluded for logistical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms as measured by the Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (CAPS-5) | Baseline, 3-months
  The CAPS-5 is a clinician-rated PTSD rating scale consisting of 30 items; the total score is calculated as the sum of 20 items assessing the 20 DSM-5 PTSD symptoms. These symptom items are scored on a 5-point scale from 0 (absent) to 4 (extreme/incapacitating). The total score of the 20 items ranges from 0 to 80 with higher scores indicating more severe PTSD symptoms. Therefore, a decrease in the total score indicates symptom improvement.

SECONDARY OUTCOMES:
Change in PTSD symptoms by the PTSD Checklist (PCL-5) | Baseline, 3-months
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses symptoms of PTSD. The PCL-5 has a variety of purposes, including monitoring symptom change during and after treatment. The minimum score is 0, the maximum is 80 (higher scores indicate increased PTSD severity).
Change in depressive symptoms measured by the Patient Health Questionnaire (PHQ-9) | Baseline, 3-months
  There are 9 questions that reflects the overall functioning and impairment due to the depressive symptoms. Scores ranges from 0 to 27, with a higher score indicating more severe symptoms.
Change in quality of life and functioning measured by the EuroQol-5 Domain (EQ-5D-5L) | Baseline, 3-months
  The EQ-5D-5L assesses patients' overall quality of life and health. This measure asks questions related to mobility, self-care, activity, pain, and anxiety/depression. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to /extreme problems. The participant indicates his/her health state by checking the box next to the most appropriate response level for each of the five dimensions. Higher scores mean better quality of life. Minimum score is 1 and the maximum score is 5 for each dimension. The measure also includes one 0-100 scale assessing how patients perceive their overall health.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Family Health Care, Baldwin, Michigan
  - Grace Health, Battle Creek, Michigan
  - Genesee Community Health Center, Flint, Michigan
  - Hamilton Community Health Network, Flint, Michigan
  - Cherry Health, Grand Rapids, Michigan
  - MidMichigan Community Health Services, Houghton Lake, Michigan
  - Upper Great Lakes Family Health Care Center, Menominee, Michigan
  - Family Medical Center of Michigan, Monroe, Michigan
  - Sterling Area Health Center, Sterling, Michigan
  - Family Care Health Centers, St Louis, Missouri
  - Western North Carolina Community Health Services, Asheville, North Carolina
  - CommUnityCare Health Centers, Austin, Texas
  - Unity Care NW, Bellingham, Washington

IPD SHARING:
Plan to Share IPD: No